CLINICAL TRIAL: NCT07174518
Title: Hormonal Impalance in Children With Simple Obesity
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ragab Hashem Abdalla, Residant doctor at Assiut university hospital, Assiut University
Other Study IDs: Hormonal impalance in obesity
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Children With Simple Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Children and adolescents aged 5 to 18 years diagnosed to be have simple obesity which it refers to excessive weight gain resulting from chronic imbalance between energy intake and energy expenditure specifically when child consumes more calories than the body uses over time with Body Mass Index (BMI) ≥ 95 th percentile on CDC growth chart

SUMMARY:
Obesity in children and adolescents is a global health issue with increasing prevalence in low and middle-income countries (LMICs) as well as a high prevalence in many high-income countries. Obesity during INTRODUCTION

childhood is likely to continue into adulthood and is associated with cardiometabolic and psychosocial comorbidity as well as premature mortality. [1] WHO defines overweight and obesity as an abnormal or excessive fat accumulation that presents a risk to health. BMI (weight/height2; kg/m2) is used as an indirect measure of body fatness in children and adolescents and should be compared with population growth references adjusted for sex and age.[2] The WHO Growth Standard is recommended in many countries for children aged 0-5 years, and for those aged 5-19 years (overweight defined as BMI ≥1SD and obesity as BMI ≥2SD of the median for age and sex), and the United States Centers for Disease Control and Prevention (CDC) Growth Reference for those aged 2 to 20 years (overweight is >85th to <95th percentile and obesity is ≥95th percentile based on CDC growth charts). [3] Abdominal or central obesity is associated with increased cardiometabolic risk in children and adolescents. For waist circumference there are regional and international growth references allowing adjustment for age and sex. A waist-to-height ratio of more than 0·5 is increasingly used as an indicator of abdominal adiposity.[4] Simple obesity, also known as primary obesity, is the most common type of obesity seen in children and adolescents. It refers to excessive weight gain resulting from a chronic imbalance between energy intake and energy expenditure, specifically when the child consumes more calories than the body uses over time.[5] Simple obesity tends to develop progressively, although it is not initially caused by endocrine dysfunction, chronic excessive adiposity may contribute to hormonal imbalances and metabolic consequences over time. These include insulin resistance, early onset of puberty, and dysregulation in the levels of key adipokines such as leptin and adiponectin. [6] It is established that excess adipose tissue can lead to significant hormonal disturbances. Adipose tissue functions as an active endocrine organ, secreting various adipokines and inflammatory mediators that disrupt normal metabolic and hormonal homeostasis.[7] One of the earliest and most critical alterations is insulin resistance, often accompanied by hyperinsulinemia. This state increases the risk of glucose intolerance and type 2 diabetes. Additionally, obese children typically exhibit leptin resistance, where elevated leptin levels fail to suppress appetite, contributing to continued weight gain. Conversely, adiponectin levels are often reduced, further impairing insulin sensitivity and promoting metabolic syndrome.[8] Obesity-related stress and inflammation can also dysregulate the hypothalamic-pituitary-adrenal (HPA) axis, leading to altered cortisol secretion, which promotes central fat accumulation and influences appetite and mood. Furthermore, obesity may affect the hypothalamic-pituitary- gonadal (HPG) axis, resulting in early puberty in girls and sometimes delayed puberty in boys, along with imbalances in sex hormones.[9]

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 5 to 18 years diagnosed to be have simple obesity which it refers to excessive weight gain resulting from chronic imbalance between energy intake and energy expenditure specifically when child consumes more calories than the body uses over time with Body Mass Index (BMI) ≥ 95 th percentile on CDC growth chart

Exclusion Criteria:

* Any obese child with:

  1. Endocrinal diseases.
  2. Syndromic obesity.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 5 to 18 years diagnosed to be have simple obesity which it refers to excessive weight gain resulting from chronic imbalance between energy intake and energy expenditure specifically when child consumes more calories than the body uses over time with Body Mass Index (BMI) ≥ 95 th percentile on CDC growth chart
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
incidance of hormonal imbalance in children with simple obesity | baseline
  evaluate hormonal imbalance in children with simple obesity